CLINICAL TRIAL: NCT02358551
Title: Comparison of Axillary Vein Puncture With Subclavian Vein Puncture in Pacemaker Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xianlun Li, Deputy Director, Department of Cardiology, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJFH-2014-086
Record Dates: First submitted 2015-01-25; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Mechanical Complication of Cardiac Pacemaker
Keywords: Pacemaker; Axillary Vein; Subclavian vein; Clinical Study; Cardiovascular implantable electronic devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axillary vein (Other): Lead Placement Through the Axillary Vein Technique
  Interventions: Device: Placement of electrode lead through axillary vein puncture
- Subclaivan vein (Other): Lead Placement Through the Subclavian Vein Technique
  Interventions: Device: Placement of electrode lead through subclavian vein puncture

INTERVENTIONS:
Device: Placement of electrode lead through axillary vein puncture
  Arms: Axillary vein
Device: Placement of electrode lead through subclavian vein puncture
  Arms: Subclaivan vein

SUMMARY:
The intrathoracic subclavian venous technique for pacemaker implantation may be associated with serious complications. Axillary vein puncture tends to reduce lead implantation complications such as pneumothorax and lead crush, but clinical adoption is not widely acknowledged, especially in China, although this approach has been proposed for 20 years. The major concern is the learning curve for axillary vein puncture and its success rate. The investigators try to prove that the success rate of axillary vein puncture is non-inferior to subclavian vein puncture, hence to promote the clinical application of axillary vein puncture to reduce pacemaker implantation complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of pacemaker or ICD implantation
* Personally signed and dated informed consent document

Exclusion Criteria:

* Accompanied with malignant disease or other disease, which cause life expectancy < 1 year.
* Anatomical variation of axillary vein or subclavian vein, unable to puncture.
* Poor compliance for follow-up.
* Patients with any condition which, in the investigator's judgment, not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of vein puncture | 1 Day

SECONDARY OUTCOMES:
Mechanical complication of electrode lead (combined endpoints of hemothorax, pneumothorax, air embolism, inadvertent arterial puncture, hematoma, fracture of electrode lead, nerve injury and subclavian crush syndrome) | 6 months
Duration of pacemaker implantation | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Xianlun Li, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

REFERENCES:
- [Derived] Liu P, Zhou YF, Yang P, Gao YS, Zhao GR, Ren SY, Li XL. Optimized Axillary Vein Technique versus Subclavian Vein Technique in Cardiovascular Implantable Electronic Device Implantation: A Randomized Controlled Study. Chin Med J (Engl). 2016 Nov 20;129(22):2647-2651. doi: 10.4103/0366-6999.193462. PMID 27823994